CLINICAL TRIAL: NCT05115955
Title: Postoperative Pain Management With Extended-release Dinalbuphine Sebacate in Patients Undergoing Arthroscopic Shoulder Surgery: a Randomized,Double-blind Study
Brief Title: PO Pain Management With Extended-release Dinalbuphine Sebacate in Patients Undergoing Arthroscopic Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chueng-He Lu, Principal Investigator, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B202105153
Record Dates: First submitted 2021-10-27; First posted 2021-11-10 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-11

CONDITIONS: Anesthesiology; Orthopedic
Keywords: Analgesia; Acute postoperative pain; Arthroscopic shoulder surgery; Randomized controlled study (RCT); Dinalbuphine sebacate; NALDEBAIN
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Control Groups; Sesame Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DS group (Experimental): Combination of routine analgesic regimen and preoperative administration of 2 ml NALDEBAIN® ER Injection (150 mg Dinalbuphine Sebacate, 75 mg/ml, 2 ml/vial).
  Interventions: Drug: DS group
- Control group (Placebo Comparator): Combination of routine analgesic regimen and preoperative administration of 2 ml sesame oil (2 ml/vial).
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: DS group — In DS group, subjects will receive intramuscular single dose of NALDEBAIN® at least 12 hours before surgery.
  Other Names: NALDEBAIN®
  Arms: DS group
Drug: Control group — In Control group, subjects will receive intramuscular 2 ml sesame oil at least 12 hours before surgery.
  Other Names: Sesame oil
  Arms: Control group

SUMMARY:
Postoperative pain is common, and the pain intensity can be moderate to severe depending on the site of surgery during the first few days after surgery, and an estimated 15% to 45% experience chronic postsurgical pain. When poorly controlled, the pain can have a significant effect on patient recovery. Proper management of postoperative pain is needed to relieve suffering and lead to earlier mobilization, shortened hospital stay, reduced hospital costs, and increased patient satisfaction. The currently proposed clinical use of Dinalbuphine Sebacate is to administer a single dose of NALDEBAIN® intramuscularly approximately 12 to 24 hours prior to the planned surgery for pain relief. Several clinical studies of NALDEBAIN® have been published, such as the use in laparotomy and laparoscopic cholecystectomy. However, toward the arthroscopic shoulder surgery, no article or report has been available publicly yet. The primary objective of this study is to determine the safety and efficacy of single doses of intramuscular NALDEBAIN® on patients scheduled to undergo arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled study. Patients scheduled to undergo arthroscopic shoulder surgery will be invited to participate in this study. After obtaining the written informed consent, each subject should be sequentially assigned an individual screening number instead of his/her name, chart number or identification. Subjects will be randomized to two groups, DS group and Control group. Both groups should be treated with both routine analgesic regimen and a dose of investigational product. Random numbers and assignment treatment were generated by computer program before this study initiated. Statistical analyses should be performed on the data to compare the two groups. Numerical variables will be present with mean and standard deviation and categorical variables will be present with number and percentage.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo arthroscopic shoulder surgery.
2. American Society of Anesthesiology Physical Class 1-3.
3. Ability and willingness to provide informed consent.

Exclusion Criteria:

1. Not willing to adhere to the study visit schedule.
2. With a history of hypersensitivity or allergy to opioids, NSAIDs or sesame oil.
3. With a medical history that may predispose them to abnormal intracranial pressure.
4. Any history of narcotic dependency, addiction, or withdrawal.
5. Any clinically significant condition that may interfere with study assessments.
6. Pregnant or breastfeeding.
7. Nonregular sinus cardiac rhythm or implanted pacemakers.
8. Prescribed antimuscarinic agents, α2-adrenergic agonists, β1-adrenergic antagonists, or antiarrhythmic agents.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Acute postoperative pain intensity | Within 1 day after surgery
  Mean pain intensity scored by numeric rating scale (NRS). Numerical Rating Scale (NRS) was a 11-point scale on which 0 represented "no pain" and 10 represented the" worst pain ever".
Brief Pain Inventory | Within 1 day after surgery
  Mean scores of each item in Brief Pain Inventory (BPI). Patients fill out 11 different NRS that ask about pain intensity and the effect of the pain on their ability to function during various activities of daily living. The severity scores range from 0 (no pain) to 10 (the most severe pain).

SECONDARY OUTCOMES:
Postoperative pain intensity | In postanesthesia care unit (PACU), and 6 hours, 7 days, 90 days, and 180 days after surgery
  Mean pain intensity scored by numeric rating scale (NRS). Numerical Rating Scale (NRS) was a 11-point scale on which 0 represented "no pain" and 10 represented the" worst pain ever".
Consumption of analgesics | Within 7 days after surgery
  The consumption of total amount (mg) of supplemental analgesics administered after surgery.
Time to the first dose of rescue medication | Up to 7 days after surgery
  Time from the end of surgery to the first rescue medication use.
Brief Pain Inventory | At baseline, 1 day, 7 days, 90 days, 180 days after surgery
  Mean scores of each item in Brief Pain Inventory (BPI). Patients fill out 11 different NRS that ask about pain intensity and the effect of the pain on their ability to function during various activities of daily living. The severity scores range from 0 (no pain) to 10 (the most severe pain).
Satisfaction assessed by a 5-point scale | 7 days after surgery
  Each subject should be asked the following question: "How satisfied were you with your post-surgical analgesia"? Subjects should be asked to classify themselves as either: 1=highly satisfied, 2=satisfied, 3=uncertain, 4=dissatisfied or 5=very dissatisfied.
Incidence of adverse events | Within 7 days after surgery
  The incidence of postoperative adverse events occurring during 7 days after surgery, especially the ones related to analgesics.

CONTACTS AND LOCATIONS:
Overall Officials: Chueng-He Lu, M.D., Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No